CLINICAL TRIAL: NCT02318732
Title: Prospective Evaluation of California's Armed and Prohibited Persons System
Brief Title: Evaluation of California's Armed and Prohibited Persons System
Acronym: APPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Rutgers University (Other); Stanford University (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 553213
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Violence
Keywords: violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): APPS intervention will be implemented in Group 1 communities prior to implementation in Group 2 communities.
  Interventions: Behavioral: APPS intervention
- Group 2 (Active Comparator): APPS intervention will be implemented in Group 2 communities following implementation in Group 1 communities.
  Interventions: Behavioral: APPS intervention

INTERVENTIONS:
Behavioral: APPS intervention — Contact with and recovery of firearms from individuals who are prohibited from possessing them

SUMMARY:
This study evaluates exposure to California's Armed and Prohibited Persons System (APPS) and risk of future violence and other important outcome events among individuals who legally purchased firearms in the past but have since become prohibited from owning them. The main hypothesis is that APPS will be associated with a significant reduction in risk for future violence among individuals who are directly affected.

DETAILED DESCRIPTION:
Violence remains an important public safety and public health problem. Prior research has shown that denying firearm purchases by individuals who are at high risk for committing violent crimes, thereby restricting their access to firearms, is an effective violence prevention strategy. The Armed and Prohibited Persons System (APPS) is a new violence prevention initiative undertaken by the California Department of Justice (CalDOJ). APPS is used by law enforcement to systematically identify persons who, having legally purchased firearms in the past, have become prohibited persons in the present-usually as the result of a criminal conviction. Such individuals are at increased risk for future violence.

APPS uses existing data to identify firearm owners among persons who have become prohibited from owning or possessing firearms under California or federal law. CalDOJ then uses this information to contact and attempt recovery of firearms in the possession of prohibited individuals.

This controlled prospective longitudinal evaluation of APPS relies principally on data collected by CalDOJ in the course of APPS operations or on data in the public domain, such as community characteristics published by the U.S. Census Bureau.

To maximize fairness during the implementation of APPS, approximately 1,000 California communities will be stratified by region, population, and violent crime rate and randomized into two groups that will be exposed to APPS at different times during the study period. Hierarchical analysis will examine outcomes for individuals clustered at the community level. The principal analysis will be on an intent to treat basis. A secondary per protocol analysis will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults with records of firearms ownership who have experienced a prohibiting event. Prohibiting events are based in Federal and California state law. Among others, they include criminal convictions for felonies and selected violent misdemeanors; emergency hospitalization for dangerousness associated with severe mental illness, as specified in statute; and status as respondent to a domestic violence restraining order.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2015-02; Primary Completion 2025-06-21 (Estimated); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of arrest for violent and firearm-related crimes | Up to 3 years
  Arrests for violent and firearm-related crimes among persons eligible for the APPS intervention

SECONDARY OUTCOMES:
Incidence of arrest for non-violent, non firearms-related crimes | Up to 3 years
  Arrests for crimes not involving violence or firearms among persons eligible for the APPS intervention
Incidence of emergency mental health hospitalizations | Up to 3 years
  Emergency mental health hospitalizations following a determination of dangerousness to self or others or grave disability among persons eligible for the APPS intervention
Incidence of domestic violence restraining orders | Up to 3 years
  Domestic violence restraining orders among persons eligible for the APPS intervention

OTHER OUTCOMES:
Community level rates of violence | Up to 3 years
  Community-level rates of violent and firearm-related crimes
Cost benefit analysis | Up to 3 years
  Assess benefits of APPS relative to costs.

CONTACTS AND LOCATIONS:
Overall Officials: Garen J Wintemute, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Sacramento, California, United States

REFERENCES:
- [Background] Wintemute GJ, Beckett L, Kass PH, Tancredi D, Studdert D, Pierce G, Braga AA, Wright MA, Cerda M. Evaluation of California's Armed and Prohibited Persons System: study protocol for a cluster-randomised trial. Inj Prev. 2017 Oct;23(5):358. doi: 10.1136/injuryprev-2016-042194. Epub 2016 Oct 11. PMID 27729440
- [Derived] Wintemute GJ, Tancredi D, Pear VA, Li Y, McCort CD, Pierce G, Braga AA, Wright MA, Laqueur H, Kravitz-Wirtz N, Studdert D, Beckett L. Population-level effects on crime of recovering firearms from armed prohibited persons: intention-to-treat analysis of a pragmatic cluster-randomised trial in California cities. Inj Prev. 2024 Oct 2:ip-2024-045234. doi: 10.1136/ip-2024-045234. Online ahead of print. PMID 39358039